ClinicalTrials.gov: NCT03599661

Principal Investigator: John M. Salsman, Ph.D.

Director of Clinical Research in Adolescent and

Young Adult Oncology

Wake Forest School of Medicine

Mollie Canzona, Ph.D.

**Co-Investigator(s):** Assistant Professor, Department of Communications

Wake Forest University

David Miller, M.D.

Professor, General Internal Medicine Epidemiology

& Prevention

Social Sciences & Health Policy Wake Forest Baptist Health

Bansari "Bonnie" Patel, M.D.

Assistant Professor, Obstetrics and Gynecology

Reproductive Medicine Wake Forest Baptist Health

Zanetta S. Lamar, M.D.

Assistant Professor, Hematology & Oncology

Comprehensive Cancer Center Wake Forest Baptis Health

**Biostatistician:** Janet A. Tooze, Ph.D.

Professor, Biostatistics

Wake Forest Baptist Comprehensive Cancer Center

**Study Coordinator:** Denisha Little-Greene, MMS

1

**Regulatory Contact:** 

Mac Robinson, PhD

Wake Forest Baptist Comprehensive Cancer Center Wake Forest University School of Medicine Medical

Protocol Editor: Center Blvd

Winston-Salem, NC 27157

Wake Forest Baptist Comprehensive Cancer Center

**Participating Institution(s):** 

**Version Date:** 06/30/2020

Amended:

Confidential

## **Table of Contents**

| 1.0 | Introduction and Background | 4 |
|---|---|---|
| 2.0 | Objectives | |
| 3.0 | Study Population | |
| 4.0 | Methods | 6 |
| 5.0 | Outcome Measures | 7 |
| 6.0 | Analytic Plan | 8 |
| 7.0 | Data Management | 9 |
| 8.0 | Confidentiality and Privacy | 9 |
| 9.0 | Data Safety and Monitoring | 10 |
| 10.0 | Reporting of Unanticipated Problems, Adverse Events or Deviations | 10 |
| Appe | ndix A – Subject Eligibility Checklist | 14 |
| Appe | ndix B – Protocol Registration Form | 14 |
| Appe | ndix C – Study Measures | 14 |

### 1.0 Introduction and Background

Every year, approximately 70,000 young adults (ages 18-39) are diagnosed with cancer, which can significantly affect their health-related quality of life in multiple areas, including the potential for infertility or other reproductive challenges. Despite this, very few young adults diagnosed with cancer are actually provided fertility preservation information let alone effective strategies or tools for how to best navigate their fertility preservation options. 1 It is critical to provide decision-making information and support about infertility risk and existing interventions to maintain reproductive potential in a delivery mode that is most congruent with this population's health communication style, such as mHealth applications. Numerous organizations, including the American Society for Reproductive Medicine (ASRM),<sup>2</sup> American Society of Clinical Oncology (ASCO),<sup>3,4</sup> and the National Comprehensive Cancer Network (NCCN),<sup>5</sup> have established national guidelines to enhance provider adherence and facilitate patient and provider discussions about fertility preservation options prior to proceeding with fertility compromising treatments. These guidelines recommend that 1) all oncologists inform their patients about the impact of their cancer and/or treatment on their fertility, and 2) all patients who solicit information about fertility preservation receive it, including a referral to a reproductive specialist when appropriate. However, previous studies suggest that oncologists face many communication challenges when discussing fertility preservation with their patients. These challenges can be related to physician attributes (e.g., knowledge barriers), patient attributes (e.g., cultural or religious prohibitions for assisted reproduction), and healthcare factors (e.g., time demands).6 In fact, a burgeoning scientific literature exists on adult oncology providers' practice patterns and barriers to discussing fertility preservation<sup>7-16</sup> and suggests that oncologists rarely refer patients to fertility preservation specialists<sup>6,10</sup> with less than 25% being aware of or distributing written educational materials to their patients<sup>10</sup> and <50% following recommended ASRM/ASCO/NCCN quidelines. 6 Similar trends hold true for the dearth of fertility preservation information and support provided to young adult cancer patients.<sup>17</sup> When more than one specialist is involved (commonly the case in young adult care), information on fertility preservation may be neglected as one specialist may assume another already discussed the topic with the patient.

Given these provider-centered obstacles, it is essential that patients can receive timely and accurate fertility preservation information via non-provider channels so they can be empowered to ask specific questions and be engaged to make appropriate decisions on their own behalf. mHealth interventions represent promising options for patient engagement, especially within a younger demographic such as young adults with cancer. Technology-enabled communications are increasingly utilized, accessible, and can be tailored to reflect specific values and preferences of a population. By delivering guideline-based fertility preservation information to young adult patients using mHealth technologies, patient knowledge may be increased and sustained, and both patients and providers may be more empowered to attend to this unaddressed issue through shared decision-making.<sup>18</sup>

This study will utilize advances in mHealth technologies to address knowledge deficits,

enhance self-efficacy, and promote shared decision-making about fertility options among newly diagnosed young adults with cancer and their providers. We will achieve this goal by developing an mHealth tool (Fertilit-e) to increase patient knowledge, thereby positively impacting self-efficacy for fertility preservation decision-making, and enhancing satisfaction with fertility preservation decisions made for this group of underserved patients. The use of mHealth interventions has grown significantly in recent years, <sup>19,20</sup> increasing the potential to make decision-making interventions more accessible, personally tailored, and integrated into clinical practice.

### 2.0 Objectives

### 2.1 Primary Objective

**2.1.1** Adapt and optimize fertility preservation content in a tailored mHealth tool for fertility preservation decision-making. More specifically, we will adapt fertility-preservation content for tailored, rapid, and clear dissemination of information in an engaging, cross-platform, patient-friendly mHealth format. We will alpha-test this tool with an ethnically diverse sample of cross-cultural end users to collect qualitative data and evaluate <u>usability</u> to refine content and design. No formal hypothesis testing will be done.

### 2.2 Secondary Objective

**2.2.1** To qualitatively evaluate comprehensibility of the mHealth tool.

## 2.3 Exploratory Objectives

- 2.3.1 To describe the characteristics of the study population in terms of health literacy, sociodemographics, technology use, and eHealth literacy.
- 2.3.2 To explore differences in usability by health literacy, sociodemographic characteristics, technology use, and eHealth literacy.

## 3.0 Study Population

Young adult patients are eligible if they: 1) are ages 18 to 39; 2) had a histologically confirmed diagnosis of cancer during ages 15 to 39, 3) will be receiving or have received treatment associated with a risk of infertility (i.e., systemic chemotherapy, pelvic radiotherapy, and/or pelvic surgery with potential impact on reproductive function), 4) considered or wish they had considered fertility preservation treatments, 5) are able to speak, read, and understand English, and 6) are able to provide electronic informed consent 7) have access to the internet 8) have access to a computer that will allow for a WebEx research interview. Young adult patients will be excluded if they: 1) had an infertility diagnosis prior to cancer diagnosis, 2) had a history of fertility preservation or fertility treatments prior to their cancer diagnosis, 3) are more than five years post-cancer-related treatments (i.e., systemic chemotherapy, pelvic radiotherapy, and/or pelvic

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

surgery). The electronic medical record will be queried to identify potentially eligible patients. IRB-approved study flyers may also be disseminated through email blasts or postings on websites of local cancer support agencies such as Cancer Services. Once potential participants have been identified, a study team member will contact patients by phone, email, and/or MyWakeHealth to describe the study, answer questions, confirm eligibility, and consent those who are interested.

Alpha testing will occur with 24 young adults. For this purposive sample, we will recruit equal numbers of men and women, one half (n=12) of our sample will be from racial or ethnic minority groups, and one fourth (n=6) will have low literacy (i.e., <12 years of education). We will recruit participants in three phases that correspond to three rounds of computer prototype testing (Round 1, n=6; Round 2, n=6; Round 3, n=12). We will strive for target representation of racial or ethnic minorities and low literacy participants within each phase.

#### 4.0 Methods

### 4.1 Registration Procedures

All patients entered on any WFBCCC trial, whether treatment, companion, or cancer control trial, **must** be linked with a study protocol in EPIC or WISER if non Wake patient within 24 hours of Informed Consent. Patients **must** be registered prior to the initiation of the study.

We will perform the following steps in order to ensure prompt registration of our patients:

- 1.0 Complete the Eligibility Checklist (Appendix A)
- 2.0 Complete the Protocol Registration Form (Appendix B)
- 3.0 Alert the Cancer Center registrar by phone, *and then* send the electronic signed Informed Consent Form, Eligibility Checklist and Protocol Registration Form to the registrar, either by fax or e-mail.

#### Contact Information:

Protocol Registrar PHONE (336) 713-6767
Protocol Registrar FAX (336) 713-6772
Protocol Registrar F MAII (registra@wakehoalth ex

Protocol Registrar E-MAIL (<u>registra@wakehealth.edu</u>)

\*Protocol Registration is open from 8:30 AM - 4:00 PM, Monday-Friday.

4.0 Fax/e-mail ALL eligibility source documents with registration. Patients **will not** be registered without all required supporting documents.

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

Note: If labs were performed at an outside institution, provide a printout of the results. Ensure that the most recent lab values are sent.

To complete the registration process, the Registrar will:

- assign a patient study number
- register the patient on the study

### 4.2 Study Procedures

Led by Dr. Miller (Co-I) and supported by Mr. Hepler (Senior Analyst and Programmer), we will configure and enable technological specifications of the alpha version of our cross platform, web-based decision-making tool. Fertilit-e will leverage the technical infrastructure from Dr. Miller's validated mPath platform (1R01CA178941), and since Fertilit-e will be web-based and cross-platform, it will be accessible across multiple different user systems and not limited to a tablet or smartphone (e.g., Android, iPhone). Further, Informed by the Ottawa Decision Support Framework, 21,22 self-efficacy theory, 23-25 and existing fertility preservation decision-aids, 26-30 we expect Fertilit-e to include, but not be limited to, the following modules: (1) personal information, values, and preferences; (2) fertility risks and options; (3) personal stories; (4) financial concerns; (5) frequently asked questions; (6) additional resources; and (7) session summary. Across all modules, the goal will be to provide tailored information (by gender) about the risks of infertility and options to preserve fertility if interested.

Alpha Testing with Patients. Aim 1 qualitative activities will be supported by the Developing Shared Resource, Q-PRO (Qualitative and Patient-Reported Outcomes) of the Wake Forest Baptist Comprehensive Cancer Center (WFBCCC). Once Fertilit-e alpha content has been developed, we will begin pilot testing the material with consented patients (n=6). Patients will meet virtually through WebEx or individually in a private setting with a member of the research team.. Participants will review a computer prototype of Fertilit-e alpha content and its design elements (see https://fertilite.phs.wakehealth.edu/). Using an interview guide (Appendix C), a research team member will ask about issues of content, functionality, and ease of use (i.e., comprehensibility and usability). Interviews will be completed within 45-60 minutes. Alpha testing will be audio and video recorded and transcripts will be de-identified prior to subsequent qualitative coding by research team member and Dr. Canzona. All participants will complete an interviewer administered screener for health literacy<sup>31,32</sup> and self-report items for technology use, eHealth literacy,33 and need for cognition.<sup>34</sup> Input will be used to modify Fertilit-e for a second round of computer prototype testing (n=6 new patients) which will follow the same process as before.

After two rounds of computer prototype testing have been completed, our

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

team will then review participant input and incorporate pertinent changes into a revised version of our decision aid that will be pilot tested with an additional 12 new patients who will use Fertilit-e on an iPad. As with earlier rounds of computer prototype testing, all participants will meet individually with a research team member in a private location. We will use the "Think Aloud" protocol to examine how individuals interact with and interpret Fertilit-e. A research team member will also ask each participant additional questions about the clarity of content and ease of use following an interview guide. At the end of alpha testing, participants will receive \$25. Feedback will be examined systematically by the study team and Advisory Board after each round of computer prototype testing to make necessary modifications prior to pilot testing in a subsequent aim.

### 5.0 Outcome Measures

### 5.1 Primary and Secondary Outcomes

To evaluate Fertilit-e alpha, we will examine its <u>comprehensibility</u> and <u>design</u> through a series of think aloud interviews<sup>35</sup> and <u>usability</u> with additional openended questions (See Appendix C). We will complement the qualitative data by administering the System Usability Scale.<sup>36,37</sup> After our alpha testing, we will have an eHealth decision aid on fertility preservation (Fertilit-e) ready to be field tested in a sample of newly diagnosed young adults with cancer.

## 6.0 Analytic Plan

### 6.1 Analysis of Primary Outcome

Q-PRO staff will review qualitative data to provide an integrative summary and identification of key points, potential themes, and areas of further exploration. A summary report will be created using the interview recordings and interviewer field notes. The report would include a summary for each module based on the data from the Think Aloud and Interview Guide that incorporates usability for Fertilit-e alpha. Q-PRO will also include a section on general comments and overall recommendations. Finally, they will be maintaining a spreadsheet that includes data for the sequence of modules selected, modules skipped, and overall time spent using the app. Q-PRO will then move to standard analysis (transcription, thematic analysis, saturation, etc.) for beta testing. <sup>38,39</sup>

Our study team will calculate descriptive statistics for the System Usability Scale by gender and race/ethnicity.

### 6.2 Analysis of Secondary Outcome

Q-PRO staff will review qualitative data that incorporates and summarizes comprehensibility for Fertilit-e alpha using the same techniques and approaches as described above (Section 6.1).

### 6.3 Analysis of Exploratory Outcomes

We will calculate descriptive statistics (means and standard deviations, frequencies) for all sociodemographic variables, the health literacy scale, 31,32 the technology use items, the eHealth literacy scale, 33 and the Need for Cognition – short form 4 to describe the study population. This will be considered exploratory due to the small sample size and intentional selection of participant groups.

To explore differences in usability by health literacy, sociodemographic characteristics, technology use and eHealth literacy, we will use t-tests, ANOVAs, and correlations to examine the relationship between these variables and the outcome of the System Usabilty Scale score.

### 6.4 Sample Size and Power

The combined sample size from each round of computer prototype testing (N=24) should permit us to achieve data saturation for gender (12 men and 12 women) With 24 participants, we will also be able to estimate the usability data within  $\pm 0.4$  SD for the System Usability Scale using 2-sided 95% confidence intervals (CIs).

#### 6.5 Accrual Rate

The WFBCCC sees a high volume of young adults with cancer annually. In the last fiscal year, 901 young adults with cancer were seen and ~550 of those were post-treatment survivors. For this purposive sampling strategy, we anticipate recruiting 24 young adults within 4 months (or 6 young adults/month). Given the relatively large sample sizes of young adults at WFBCCC, we believe our proposed sample sizes and timeline are realistic goals.

### 6.6 Length of Study

Patients will complete their participation in 45-60 minutes. We expect the entire qualitative data collection will be completed within 4 months.

## 7.0 Data Management

| Informed consent document | EPIC/REDCap |
|----------------------------|--------------|
| Protocol registration form | WISER/OnCore |
| Study questionnaire | REDCap |

## 8.0 Confidentiality and Privacy

Confidentiality will be protected by collecting only information needed to assess study outcomes, minimizing to the fullest extent possible the collection of any information that could directly identify subjects, and maintaining all study information in a secure manner. To help ensure subject privacy and confidentiality, only a unique study identifier will appear on the data collection form. Any collected patient identifying information corresponding to the unique study identifier will be maintained on a linkage

file, store separately from the data. The linkage file will be kept secure, with access limited to designated study personnel. Following data collection, subject identifying information will be destroyed, consistent with data validation and study design, producing an anonymous analytical data set. Data access will be limited to study staff. Data and records will be kept locked and secured, with any computer data password protected. No reference to any individual participant will appear in reports, presentations, or publications that may arise from the study.

### 9.0 Data Safety and Monitoring

The principal investigator will be responsible for the overall monitoring of the data and safety of study participants. The principal investigator will be assisted by other members of the study staff.

The risks of this study are low; however, staff will be trained to handle situations with sensitivity and empathy. The study coordinator will be trained to monitor for significant patient distress or depressive symptoms and will be instructed on the appropriate courses of referral is a patient is considered to be at risk for a safety concern.

## 10.0 Reporting of Unanticipated Problems, Adverse Events or Deviations

Any unanticipated problems, serious and unexpected adverse events, deviations or protocol changes will be promptly reported by the principal investigator or designated member of the research team to the IRB and sponsor or appropriate government agency if appropriate.

In the rare event that a participant becomes distressed as a result of participating in this study or rather becomes more reflective and wants to talk about these issues in more depth, we will provide referrals to members of the psychosocial support team and/or other clinical staff as appropriate.

#### References

- Clayman ML, Harper MM, Quinn GP, Reinecke J, Shah S. Oncofertility Resources at NCI-Designated Comprehensive Cancer Centers. J Natl Compr Canc Netw. 2013;11(12):1504-1509.
- 2. Ethics Committee of the American Society for Reproductive Medicine. Fertility preservation and reproduction in cancer patients. *Fertil Steril.* 2005;83(6):1622-1628.
- 3. Lee SJ, Schover LR, Partridge AH, et al. American Society of Clinical Oncology recommendations on fertility preservation in cancer patients. *J Clin Oncol*. 2006;24(18):2917-2931.
- 4. Loren AW, Mangu PB, Beck LN, et al. Fertility Preservation for Patients With Cancer: American Society of Clinical Oncology Clinical Practice Guideline Update. *J Clin Oncol.* 2013;31(19):2500-2510.
- 5. Coccia PF, Altman J, Bhatia S, et al. Adolescent and young adult oncology clinical practice guidelines in oncology. *J Natl Compr Canc Netw.* 2012;10(9):1112-1150.
- 6. Knapp CA, Quinn GP. Healthcare provider perspectives on fertility preservation for cancer patients. *Cancer Treat Res.* 2010;156:391-401.
- 7. King L, Quinn GP, Vadaparampil ST, et al. Oncology nurses' perceptions of barriers to discussion of fertility preservation with patients with cancer. *Clin J Oncol Nurs*. 2008;12(3):467-476.
- 8. Quinn G, Vadaparampil S, Gwede C, et al. Discussion of fertility preservation with newly diagnosed patients: oncologists' views. *J Cancer Surviv.* 2007;1(2):146-155.
- 9. Quinn GP, Murphy D, Knapp C, et al. Who Decides? Decision Making and Fertility Preservation in Teens With Cancer: A Review of the Literature. *J Adolesc Health*. 2011;49(4):337-346.
- 10. Quinn GP, Vadaparampil ST. Fertility Preservation and Adolescent/Young Adult Cancer Patients: Physician Communication Challenges. *J Adolesc Health*. 2009;44(4):394-400.
- 11. Quinn GP, Vadaparampil ST, Gwede CK, Bell-Ellison BA, Albrecht TL. Patient-physician communication barriers regarding fertility preservation among newly diagnosed cancer patients. *Soc Sci Med.* 2008;66(3):784-789.
- 12. Quinn GP, Vadaparampil ST, Gwede CK, Mason TM, Reinecke JD, Silva C. Developing a referral system for fertility preservation among patients with newly diagnosed cancer. *J Natl Compr Canc Netw.* 2011;9(11):1219-1225.
- 13. Quinn GP, Vadaparampil ST, King L, et al. Impact of physicians' personal discomfort and patient prognosis on discussion of fertility preservation with young cancer patients. *Patient Educ Couns.* 2009;77(3):338-343.
- 14. Quinn GP, Vadaparampil ST, Lee JH, et al. Physician referral for fertility preservation in oncology patients: A national study of practice behaviors. *J Clin Oncol.* 2009;27(35):5952-5957.

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

- 15. Clayton H, Quinn GP, Lee JH, et al. Trends in clinical practice and nurses' attitudes about fertility preservation for pediatric patients with cancer. *Oncol Nurs Forum.* 2008;35(2):249-255.
- Schover LR, Brey K, Lichtin A, Lipshultz LI, Jeha S. Oncologists' attitudes and practices regarding banking sperm before cancer treatment. *J Clin Oncol*. 2002;20(7):1890-1897.
- 17. Clayman M, Arntson P, Galvin K. Shared decision making: Fertility and pediatric cancers. In: Woodruff TK, Snyder KA, eds. *Oncofertility fertility preservation for cancer survivors*. New York: Springer Verlag; 2007:149-160.
- 18. Knapp CA, Quinn GP. Healthcare provider perspectives on fertility preservation for cancer patients. In: Woodruff TK, ed. *Oncofertility: ethical, legal, social, and medical perspectives.* New York: Springer; 2010:391-401.
- 19. Demiris G, Afrin LB, Speedie S, et al. Patient-centered applications: use of information technology to promote disease management and wellness. A white paper by the AMIA knowledge in motion working group. *J Am Med InformAssoc*. 2008;15(1):8-13.
- 20. Glasgow RE, Davis CL, Funnell MM, Beck A. Implementing practical interventions to support chronic illness self-management. *JtComm J Qual Saf.* 2003;29(11):563-574.
- 21. O'Connor AM, Drake ER, Fiset V, Graham ID, Laupacis A, Tugwell P. The Ottawa patient decision aids. *Eff Clin Pract*. 1999;2(4):163-170.
- 22. O'Connor AM, Jacobsen MJ, Stacey D. An evidence-based approach to managing women's decisional conflict. *J Obstet Gynecol Neonatal Nurs.* 2002;31(5):570-581.
- 23. Bandura A. Self-efficacy: Toward a unifying theory of behavioral change. *Psychol Rev.* 1977;84(2):191-215.
- 24. Bandura A. Self-efficacy mechanism in human agency. *Am Psychol.* 1982;37(2):122-147.
- 25. Bandura A. *Self-efficacy: the exercise of control.* New York: W.H. Freeman; 1997.
- 26. Block R, Nail L, Frohnmayer A, et al. The Fertility Preservation Explorer: A Decision Tool for Adolescent and Young Adult Women with Cancer. Paper presented at: Oncofertility Consortium 2013; Chicago, IL.
- 27. Block R, Nail L, Frohnmayer A, Hayes-Lattin B. The fertility preservation decision-making process of adolescent and young adult women with cancer. Paper presented at: International Society of Pediatric Oncology (SIOP) October 28-30, 2011; Auckland, New Zealand.
- 28. Northwestern University. myoncofertility.org. 2011; <a href="http://www.myoncofertility.org/">http://www.myoncofertility.org/</a>. Accessed February 1, 2014.
- 29. Northwestern University. Patient Navigator for Fertility Preservation. 2011; <a href="http://fertilitypreservation.northwestern.edu/">http://fertilitypreservation.northwestern.edu/</a>. Accessed February 1, 2014.
- 30. Northwestern University. iSaveFertility iOS Application. 2011; <a href="https://itunes.apple.com/us/app/isavefertility/id436397171?mt=8&ls=1">https://itunes.apple.com/us/app/isavefertility/id436397171?mt=8&ls=1</a>.
- 31. Chew LD, Griffin JM, Partin MR, et al. Validation of screening questions for limited health literacy in a large VA outpatient population. *J Gen Intern Med.* 2008;23(5):561-566.

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

- 32. Wallston KA, Cawthon C, McNaughton CD, Rothman RL, Osborn CY, Kripalani S. Psychometric properties of the brief health literacy screen in clinical practice. *J Gen Intern Med.* 2014;29(1):119-126.
- 33. Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. *J Med Internet Res.* 2006;8(4):e27.
- 34. Cacioppo JT, Petty RE, Kao CF. The efficient assessment of need for cognition. *J Pers Assess.* 1984;48(3):306-307.
- 35. Kelly-Blake K, Clark S, Dontje K, et al. Refining a brief decision aid in stable CAD: cognitive audios. *BMC Med Inform Decis Mak.* 2014;14(1):10.
- 36. Brooke J. SUS-A quick and dirty usability scale. *Usability evaluation in industry*. 1996;189(194):4-7.
- 37. Bangor A, Kortum PT, Miller JT. An Empirical Evaluation of the System Usability Scale. *Int J Hum Comput Interact.* 2008;24(6):574-594.
- 38. Bowen GA. Naturalistic inquiry and the saturation concept: a research note. *Qual Res.* 2008;8(1):137-152.
- 39. Guest G, Bunce A, Johnson L. How Many Interviews Are Enough? An Experiment with Data Saturation and Variability. *Field Meth.* 2006;18(1):59-82.

## Appendix A – Subject Eligibility Checklist

| IRB Protocol No. | | \ | WFBCCC Protocol No |
|---|---|---|---|
| Study Title: Fertilit-e | | | |
| Principal Investigator: John M. Salsman | n, Ph.D. | | |
| Inclusion Criteria (as outlined in study protocol) | Criteria<br>is met | Criteri<br>is NO<br>met | |
| Age 18 to 39. | | | |
| Histologically confirmed diagnosis of cancer during ages 15 to 39 | | | |
| Will be receiving or have received treatment associated with a risk of infertility (i.e., chemotherapy, pelvic radiotherapy, and/or pelvic surgery with potential impact on reproductive function). | | | |
| Considered or wish they had considered fertility preservation treatments. | | | |
| Able to speak, read, and understand English. | | | |
| Able to provide informed consent. | | | |
| Have internet access | | | |
| Have a laptop, or desktop computer that can connect to WebEx | | | |
| Exclusion Criteria (as outlined in study protocol) | Criteria<br>NOT<br>present | Criteri<br>is<br>presei | (Please document dates and lab |
| Infertility diagnosis prior to cancer diagnosis. | | | |
| History of fertility preservation or fertility treatments prior to their cancer diagnosis. | | | |
| Are more than five years post-cancer-<br>related treatments (i.e., systemic<br>chemotherapy, pelvic radiotherapy,<br>and/or pelvic surgery) | | | |
| This subject is eligible / ineligible for participation in this study. | | | |
| OnCore Assigned PID: | | | |
| Signature of research professional confirming eligibility: | | | |
| Date: // | | | |

| Signature of Treating Physician* | k | |
|---|---|---|
| laboratory results, etc. When listing | the source, spec<br>nclude the date o | urce documents include clinic note, pathology report, ifically state which document in the medical record on the document. Example: "Pathology report, lowing registration if needed |
| Appendix B– Reduced F | Review** Re | gistration Form |
| DEMOGRAPHICS | | |
| Patient: Last Name: | | First Name: |
| MRN: | | ZIPCODE: |
| *SEX: □ Male □ Fem | ale | |
| *Ethnicity (choose one): | □ Hispanic | □Non-Hispanic |
| *Race (choose all that apply): | □ WHITE | □African American |
| | ☐ ASIAN | ☐ PACIFIC ISLANDER |
| | □ NATIVE A | MERICAN (Alaskan) |
| *Diagnosis: | | |
| DOB (mm/dd/yy): // | / | (include if no MRN is provided) |
| *MD Name (Last, First) : | | <u> </u> |
| *Date Consent Signed: | - | |
| Date of Registration: (if different | Date of Registration: (if different than | |
| consent signing) | | |
| PID # (OnCore): | | (to be completed by registrar) |

The Comprehensive Cancer Center requires that all registrations be sent to the CCCWFU Centralized Registrar the day the patient is consented; if this is not possible we require that all registration be communicated to the Centralized Registrar within 72 hours by the CRM registrar.

For questions, the Protocol Registrar can be contact by calling 336-713-6767 between 8:30 AM and 4:00 PM, Monday – Friday.

Completed Eligibility Checklist and Protocol Registration Form must be hand delivered, faxed or e-mailed to the registrar at 336-713-6772 or <a href="registra@wakehealth.edu">registra@wakehealth.edu</a>.

<sup>\*\*</sup>Reduced Review means eligibility and other review are not performed by CRM registrar.

\*\*\* if not using the full wakehealth.edu outlook client (full outlook, not web outlook) save this file and attach to an email to <a href="mailto:registra@wakehealth.edu">registra@wakehealth.edu</a>.

Submitter of this form is responsible for insuring that all regulatory and eligibility requirements are met for this registration

### **APPENDIX C. Data Collection Measures**

| Variable/Construct | Measure | Items | Source |
|---|---|---|---|
| Health Literacy | Brief Health Literacy Screener | 3 | Chew et al., 2008; |
| | | | Wallston et al., 2014 |
| Patient | Sociodemographic variables | 23 | Standard items |
| Characteristics | | | |
| Technology Use | Type, frequency, and purpose | 11 | Study team developed |
| | of technology use variables | | |
| eHealth Literacy | Questions about comfort with | 10 | Norman & Skinner, |
| | and use of eHealth information | | 2006 |
| Need for Cognition | Need for Cognition Scale | 18 | Cacioppo et al., 1984 |
| Comprehensibility | Interview Guide | 10 | Study team developed |
| | | | and informed by Kelly- |
| | | | Blake et al., 2014 |
| Usability | Interview Guide; | 11; | study team developed; |
| | System Usability Scale | 12 | Brooke, 1996 |

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

## BRIEF HEALTH LITERACY SCREENER

| 1. | How often do you have someone (like a family member, friend, hospital/clinic worker of caregiver) help you read hospital materials? (Help Read) all of the time some of the time a little of the time none of the time Refused [DO NOT READ] |
|---|---|
| 2. | How often do you have problems learning about your medical condition because of difficulty understanding written information? (Problems Learning), all of the time most of the time a little of the time none of the time Refused [DO NOT READ] |
| 3. | How confident are you filling out medical forms by yourself? (Confident with Forms) cut extremely cut a bit somewhat a little bit not at all Refused [DO NOT READ] |

Chew LD, Griffin JM, Partin MR, et al. Validation of screening questions for limited health literacy in a large VA outpatient population. *J Gen Intern Med.* 2008;23(5):561-566.

Wallston KA, Cawthon C, McNaughton CD, Rothman RL, Osborn CY, Kripalani S. Psychometric properties of the brief health literacy screen in clinical practice. *J Gen Intern Med*. 2014;29(1):119-126.

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

### Patient Sociodemographic Variables

This set of questions is about your cancer treatment and general background. Unless otherwise stated, please select only one response for each question. All of the information you provide is confidential.

| What | is your current cancer treatment plan? Check all that apply |
|--------|-------------------------------------------------------------|
| | I have not had any treatment |
| | I am currently receiving chemotherapy |
| | I am currently receiving radiation |
| | I have had surgery to remove or treat cancer or tumor |
| | I have completed treatment |
| | Other (please describe:) |
| What | is your gender? |
| | Male |
| | Female |
| | Transgender |
| | Tunigender |
| • | ou of Hispanic, Latino, or Spanish origin or descent? |
| | Yes, Hispanic, Latino, or Spanish |
| Ц | No, not Hispanic, Latino, or Spanish |
| What | is your race? (check all that apply) |
| | White |
| | Black or African American |
| | Asian |
| П | Native Hawaiian or Other Pacific Islander |
| | American Indian or Alaska Native |
| | Other |
| What i | s your residential zip code? |
| What | is your present religion, if any? |
| | Protestant; if yes, which denomination? |
| | Roman Catholic |
| | Mormon |
| | Orthodox such as Greek or Russian Orthodox |
| | Jewish |
| | Muslim |
| | Buddhist |
| | Hindu |
| | Atheist |
| | Agnostic |
| | Other |
| | No particular religion |

# Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717 tant are your religious or spiritual beliefs to you?

| | mportant are your religious or spiritual beliefs to you? |
|---|---|
| | Not at all |
| | A little bit |
| | Somewhat |
| | Quite a bit |
| | Very much |
| What | is the highest grade or level of school that you have completed? |
| | 8th grade or less |
| | Some high school, but did not graduate |
| | High school graduate or GED |
| | Some college or 2-year degree |
| | 4-year college graduate |
| | More than 4-year college degree |
| What | was your employment or school status <u>JUST BEFORE</u> your cancer diagnosis? |
| (check | x all that apply): |
| | Employed full-time (including self-employed) |
| | Employed part-time (including self-employed) |
| | Full-time homemaker |
| | Full-time student |
| | On temporary medical leave/disability |
| | Unemployed |
| | Permanently unable to work |
| What | is your employment or school status <b>NOW</b> ? (check all that apply): |
| | Employed full-time (including self-employed) |
| | Employed part-time (including self-employed) |
| | Full-time homemaker |
| | Full-time student |
| | On temporary medical leave/disability |
| | Unemployed |
| | Permanently unable to work |
| | is your current marital / relationship status? |
| | Single / Never married |
| | Single/Divorced |
| | Single/Widowed |
| | Married or living with partner in committed relationship |
| | Married but currently separated |
| Who l | ives at home with you? (check all that apply): |
| | Parent(s) |
| | Grandparents |
| | Siblings |
| | Spouse |

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

| | Significant other/partner Child(ren) Number of children Friend(s)/Roommate(s) I live alone Other, please specify |
|---|---|
| | Me My spouse or significant other My child My parent(s)* [If patient selects this option, please skip to "In general, would you say your health is" item.] Someone else not listed here, please specify There is no income earner in my household |
| housel | None 1 2 3 |
| yourse | the categories below, please indicate the annual income of your household. Include elf and anyone you live and share finances with. Less than \$15,000 \$15,000 to \$29,999 \$30,000 to \$59,999 \$60,000 to \$100,000 More than \$100,000 Do not know |
| | No No, but I have applied for disability Yes, short term disability (i.e., pays you a portion of your income for a short period of time after you run out of sick leave; depending on your plan, it will generally pay you for between 9 and 52 weeks) Yes, long term disability (i.e., pays you a portion of your income after you run out of both sick leave and short term disability, Social Security Disability Insurance or Supplemental Security Income) Yes, I am permanently disabled |

What is your current primary health insurance provider (mark one)

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

| <ul> <li>☐ Me</li> <li>☐ Pri</li> <li>☐ Ve</li> </ul> | alified health plan from the Health Insurance Marketplace |
|---|---|
| □ No<br>□ Yes | |
| ☐ Exc | ry good<br>ood<br>ir |
| How man | y biological children do you have? |
| ☐ Fer☐ I do☐ I'm☐ I'm | ou feel about preserving your fertility right now? rtility preservation is not for me. I'm here to learn about my options just in case. on't think fertility preservation is right for me. I don't know if there is a good option. n not sure about what to do. I want to explore my options. n interested in fertility preservation. I want to compare my options. vant to preserve my fertility. I am ready to select a method. |
| ☐ Ven☐ Qu☐ Son☐ A l | awareness of treatments to protect your ability to become a parent ry much ite a bit mewhat little bit at all |
| ☐ Ven☐ Qu☐ Son | comfort level with treatments to protect your ability to become a parent ry much ite a bit mewhat little bit at all |
| ☐ Yes | obably yes |

| Wake Forest Baptist Comprehensive Cancer Center (WFBCCC |
|---------------------------------------------------------|
| WFBCCC # 01717 |
| Probably no |
| No |

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

## The next set of questions will ask you about your use of technology.

| | u have a cellphone? Yes – a cellphone Yes – a smartphone No |
|---|---|
| | Property is the second of the |
| | you used a computer or laptop in the last 30 days? Yes No |
| | u have a computer or laptop that you could use in your home? Yes No |
| | u use the internet?<br>Yes<br>No |
| On a s | How often do you access the internet? smartphone Every day or almost every day 3 to 5 days a week 1 to 2 days a week Once or twice a month Less than once a month Never |
| | Every day or almost every day 3 to 5 days a week 1 to 2 days a week Once or twice a month Less than once a month Never |
| | aptop or computer Every day or almost every day |

| | WFBCCC # 01/1/ |
|---|---|
| | 3 to 5 days a week |
| | 1 to 2 days a week |
| | Once or twice a month |
| | Less than once a month |
| | Never |
| | of the following sources did you use to get information about cancer-related dity and treatment options to preserve fertility? (choose all that apply) |
| | Physicians |
| | Nurses |
| | Family and friends |
| | Books/magazines |
| | E |
| | Internet |
| | of the following statements best describes your preferred approach to making al decisions: (please choose only <u>one</u> answer) |
| | I prefer to make the final decision about which treatment I will receive. |
| | • |
| | doctor's opinion |
| | I prefer that my doctor and I share responsibility for deciding which treatment is best for |
| | me. I made that may do ston makes the final decision about which treatment will be used but |
| | I prefer that my doctor makes the final decision about which treatment will be used, but seriously considers my opinion. |
| | I prefer to leave all decisions regarding treatment to my doctor. |
| | I prefer to feave an decisions regarding treatment to my doctor. |
| | of the following best describes the role you played when the decision was made treatment for your cancer-related infertility? (please choose only <u>one</u> answer) |
| | I made the final decision about which treatment I received. |
| | I made the final decision about my treatment after seriously considering my doctor's opinion |
| | My doctor and I shared responsibility for deciding which treatment was best for me. |
| | My doctor made the final decision about which treatment would be used, but seriously |
| | considered my opinion. My doctor made all treatment decisions |
| _ | , |

#### eHealth Literacy Scale

The following questions are about your opinion and experiences using the internet for health information. For each statement, tell me which response best reflects your opinion and experience *right now*.

1. How **useful** do you feel the Internet is in helping you in making decisions about your health?

| <b>□</b> 1 | П2 | □3 | □4 | □5 |
|-------------------|------------|--------|--------|-------------|
| Not useful at all | Not useful | Unsure | Useful | Very Useful |

2. How **important** is it for you to be able to access health resources on the Internet?

| <b>□</b> 1 | □2 | □3 | □4 | □5 |
|---|---|---|---|---|
| Not<br>important<br>at all | Not important | Unsure | Important | Very<br>important |

| 2 | I know what | health rec | Olltoge ara | availabla | on the | Internet |
|---|---|---|---|---|---|---|
| • | i know <b>wnat</b> | nealth res | ources are | avanable | on the | ınremer |

- 1) ☐ Strongly Disagree
- 2) ☐ Disagree
- 3) □ Undecided
- 4) ☐ Agree
- 5) ☐ Strongly Agree

4. I know **where** to find helpful health resources on the Internet.

- 1) ☐ Strongly Disagree
- 2) □ Disagree
- 3) □ Undecided
- 4) ☐ Agree
- 5) ☐ Strongly Agree

5. I know **how** to find helpful health resources on the Internet.

- 1) ☐ Strongly Disagree
- 2) ☐ Disagree
- 3) □ Undecided
- 4) ☐ Agree

| 5) LI Strongly Agree |
|---|
| 6. I know <b>how to use</b> the Internet to answer my questions about health. |
| 1) □ Strongly Disagree |
| 2) □ Disagree |
| 3) □ Undecided |
| 4) □ Agree |
| 5) □ Strongly Agree |
| 7. I know how to use <b>the health information</b> I find on the Internet to help me. |
| 1) ☐ Strongly Disagree |
| 2) □ Disagree |
| 3) □ Undecided |
| 4) □ Agree |
| 5) □ Strongly Agree |
| 8. I have the skills I need to <b>evaluate</b> the health resources I find on the Internet. |
| 1) □ Strongly Disagree |
| 2) □ Disagree |
| 3) □ Undecided |
| 4) □ Agree |
| 5) □ Strongly Agree |
| 9. I can tell <b>high quality</b> health resources from <b>low quality</b> health resources on the Internet |
| 1) □ Strongly Disagree |
| 2) □ Disagree |
| 3) □ Undecided |
| 4) □ Agree |
| 5) □ Strongly Agree |
| 10. I feel <b>confident</b> in using information from the Internet to make health decisions. |
| 1) □ Strongly Disagree |
| 2) □ Disagree |
| 3) □ Undecided |
| 4) □ Agree |
| 5) □ Strongly Agree |

## Wake Forest Baptist Comprehensive Cancer Center (WFBCCC) WFBCCC # 01717

#### Need for Cognition Scale (from Cacioppo, Petty, & Kao, 1984)

For each of the statements below, please indicate whether or not the statement is characteristic of you or of what you believe. For example, if the statement is extremely uncharacteristic of you or of what you believe about yourself (not at all like you) please place a "1" on the line to the left of the statement. If the statement is extremely characteristic of you or of what you believe about yourself (very much like you) please place a "5" on the line to the left of the statement. You should use the following scale as you rate each of the statements below.

| extremely<br>uncharacteristic<br>of me | | somewhat<br>uncharacteristic<br>of me | uncertain | somewhat characteristic of me | extremely<br>characteris<br>of me |
|---|---|---|---|---|---|
| 1 | l wou | ld prefer complex to | simple proble | ems. | |
| 2 | I like t | to have the responsi | bility of handl | ing a situation that | requires a lot of |
| 3 | | ing is not my idea of | ffun.** | | |
| 4 | | ld rather do somethi<br>s sure to challenge n | • | uires little thought than something abilities.** | |
| 5 | • | o anticipate and avoi<br>to think in depth abo | | | ely chance I will |
| 6 | I find | satisfaction in delibe | erating hard a | nd for long hours. | |
| 7 | I only think as hard as I have to.** | | | | |
| 8 | I prefe | er to think about sma | all daily projec | ets to long term one | ?S.** |
| 9 | l like t | tasks that require litt | le thought one | ce I've learned ther | n.** |
| 10 | The id | dea of relying on tho | ught to make | my way to the top | appeals to me. |
| 11 | I really enjoy a task that involves coming up with new solutions to p | | | | |
| 12 | Learning new ways to think doesn't excite me very much.** | | | | |
| 13 | I prefer my life to be filled with puzzles I must solve. | | | | |
| 14. | The n | otion of thinking abs | stractly is appe | ealing to me. | |

| 15 | I would prefer a task that is intellectual, difficult, and important to one that is somewhat important but does not require much thought. |
|---|---|
| 16 | I feel relief rather than satisfaction after completing a task that requires a lot of mental effort.** |
| 17 | It's enough for me that something gets the job done; I don't care how or why it works.** |
| 18 | I usually end up deliberating about issues even when they do not affect me personally. |

Note: \*\*=reverse scored item.

### Please see IRB for Fertilit-e Alpha Testing Interview Guide 8.27.18

### **System Usability Scale**

For the next questions, please read each sentence and rate your level of agreement.

| | | Strongly<br>disagree | | | | Strongly<br>agree |
|---|---|---|---|---|---|---|
| 1 | I think that I would like to use<br>Fertilit-e frequently (when<br>thinking about my fertility<br>options) | 1 | 2 | 3 | 4 | 5 |
| 2 | I found Fertilit-e unnecessarily complex | 1 | 2 | 3 | 4 | 5 |
| 3 | I thought Fertilit-e was easy to use | 1 | 2 | 3 | 4 | 5 |
| 4 | I think that I would need the support of a technical person to be able to use Fertilit-e | 1 | 2 | 3 | 4 | 5 |
| 5 | I found the various functions in Fertilit-e were well integrated | 1 | 2 | 3 | 4 | 5 |
| 6 | I thought there was too much inconsistency in Fertilit-e | 1 | 2 | 3 | 4 | 5 |
| 7 | I would imagine that most people would learn to use Fertilit-e very quickly | 1 | 2 | 3 | 4 | 5 |
| 8 | I found Fertilit-e very cumbersome to use | 1 | 2 | 3 | 4 | 5 |
| 9 | I felt very confident using Fertilit-e | 1 | 2 | 3 | 4 | 5 |
| 10 | I needed to learn a lot of<br>things before I could get going<br>with Fertilit-e | 1 | 2 | 3 | 4 | 5 |
| 11 | Compared to reading a brochure, I liked using Fertilit-e more. | 1 | 2 | 3 | 4 | 5 |

| 12. O | verall, would you rate the user-friendliness of Fertilit-e as: |
|-------|----------------------------------------------------------------|
| | Excellent |
| | Good |
| | OK |
| | Poor |
| | Δwful |

Brooke J. SUS-A quick and dirty usability scale. Usability evaluation in industry. 1996;189(194):4-7.